CLINICAL TRIAL: NCT01907750
Title: Transcystic Versus Transanastomotic Biliary Drainage Tubes in Living Donor Liver Transplantation. A Prospective Randomized Trial.
Brief Title: Transcystic Versus Transanastomotic Tube Drainage in Right Lobe LDLT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Ahmad Sultan, Assistant professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Biliary_TCvsTA
Record Dates: First submitted 2013-06-23; First posted 2013-07-25 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Living Donor Liver Transplantation
Keywords: biliary fistula; biliary stricture; biliary drainage tube
MeSH Terms: conditions — Biliary Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transanastomotic tube (Active Comparator): use of transanastomotic tube.
  Interventions: Device: biliary drainage tube
- Transcystic tube (Active Comparator): use of transcystic tube to drain bile duct
  Interventions: Device: biliary drainage tube

INTERVENTIONS:
Device: biliary drainage tube

SUMMARY:
To evaluate the safety and effectiveness of the use of transcystic biliary drainage tube (not transanastomotic) in comparison to the usual transanastomotic biliary drainage tube.

DETAILED DESCRIPTION:
a biliary drainage tube is usually inserted into the biliary passage after choledocho-choledochostomy (bile duct to bile duct joining).

A 4F or 5F biliary catheter (Marquat Genie biomedical, france) is used in all cases.

the study is to compare the effectiveness and safety of 2 different placement techniques:

1. the usual trans-anastomotic position (the tube is placed across the anastomosis line with the tip inside the intrahepatic biliary branches) through an opening in the wall of the recipient's common bile duct
2. a transcystic non-anastomotic position (the tube is placed through the cystic duct opening into the distal common bile duct not passing through anastomosis)

ELIGIBILITY:
Inclusion Criteria:

* living donor liver transplantation
* single bile duct in the graft

Exclusion Criteria:

* multiple bile ducts

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-01; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
early postoperative biliary fistula | 2 weeks

SECONDARY OUTCOMES:
biliary stricture | 2 years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M Sultan, MD, PhD, Principal Investigator — Gastro-enterology surgical center, Mansoura University; Mohammed Abdul-Wahab, MD, PhD, Study Chair — Gastro-enterolgy surgical center, Mansoura University; Tarek Salah, MD, PhD, Study Director — Gastro-enterolgy surgical center, Mansoura University
Locations (1):
- Gastro-enterolgy surgical center, Mansoura University, Al Mansurah, Al-Dakahleia, Egypt